CLINICAL TRIAL: NCT04413721
Title: Effects of Packed Red Blood Cell Storage Duration on Pediatric Living Donor Liver
Brief Title: Effects of Packed Red Blood Cell Storage Duration on Pediatric Living Donor Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Dr., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBC20200505
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Transfusion Related Complication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term storage RBCs (stored for ≤ 14 days) (Experimental): patients in this group were transfused with short-term storage RBCs (stored for ≤ 14 days).
  Interventions: Procedure: RBC transfustion
- Longer-term storage RBCs (stored for ≥21 days) (Active Comparator): patients in this group were transfused with longer-term storage RBCs (stored for ≥21 days).
  Interventions: Procedure: RBC transfustion

INTERVENTIONS:
Procedure: RBC transfustion — When the hemoglobin concentration fell below 7.0 g per deciliter, RBC were given to maintain the hemoglobin concentrations in the range of 7.0 to 10.0g /dL

SUMMARY:
The patients assigned to either short-storage leukoreduced RBCs group (stored for ≤ 14 days) or longer-term storage leukoreduced RBCs group(stored for ≥21 days).When the hemoglobin concentration fell below 7.0 g per deciliter, PRBC were given to maintain the hemoglobin concentrations in the range of 7.0 to 10.0/dL. The primary outcome : Death from all causes in1-year after randomization. Secondary outcomes included: Intraoperative blood transfusion, Postoperative blood transfusion, Postoperative inflammatory reaction, Mechanical ventilation time in the intensive care unit, Lengths of stay in the intensive care unit and the hospital were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Our study included pediatric patients (6 months< the moon's age <36 months) who will receive standard living-donor liver transplantation (LDLT) in Renji Hospital.

Exclusion Criteria:

* The exclu¬sion criteria of the study were a congenital sufferer from heart, lung, kidney, nervous system or blood disease,active Lung infection，a history of liver transplantation，Multivisceral transplantation , refused to participate the study.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality in in1-year after randomization | 1-year after randomization.
  Death from all causes in1-year after randomization.